CLINICAL TRIAL: NCT04218669
Title: A Clinical Randomized Trial Comparing T-tube Drainage Versus Choledochojejunostomy in Hepatolithiasis Patients With Sphincter of Oddi Laxity
Brief Title: The Approach of Biliary Drainage in Hepatolithiasis Patients With Sphincter of Oddi Laxity
Acronym: BD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: xpgeng (Other)
Responsible Party: Sponsor-Investigator, xpgeng, professor, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1804h08020239
Record Dates: First submitted 2019-12-31; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Sphincter of Oddi Laxity
Keywords: sphincter of Oddi laxity; hepatolithiasis; choledochojejunostomy

STUDY DESIGN:
Intervention Model Description: Patients were randomized to choledochojejunostomy arm or T tube drainage arm
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the surgeons and patients is not feasible due to the obviously different characteristics of the two types of biliary drainage.
  Investigator and outcome assessors will be blinded to the trial intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-tube drainage (Active Comparator): The T-tube was placed for biliary drainage
  Interventions: Procedure: T-tube drainage
- Roux-en-Y Hepaticojejunostomy (Experimental): biliary-enteric anastomosis was performed
  Interventions: Procedure: Roux-en-Y Hepaticojejunostomy

INTERVENTIONS:
Procedure: Roux-en-Y Hepaticojejunostomy — The common hepatic duct was cut and the duodenal side is closed by suture. The small intestine was cut off 15 cm below the ligament of Treitz. The distal end was lifted, and a 1-2 cm incision was made at the jejunal wall 4-5 cm from the jejunal stump. The anastomosis is used a 5-0 PSD Ⅱ suture, with double needles, inside-out in the jejunum and outside-in in the hepatic duct. One side of needles was used to continuely penetrate and suture the whole layer of the posterior-lateral wall of the jejunum, the posterior-lateral wall of the biliary duct, and the other side of needles was used to continuely stuere the anterior part of the anastomosis. Mucosa-to-mucosa contact should be ensured with every stitch.The anastomotic stomas were then checked for leakage. Enteric-enteric anastomosis was performed 60 cm below the site of the hepatojejunal anastomosis.
  Arms: Roux-en-Y Hepaticojejunostomy
Procedure: T-tube drainage — The T-tube was placed for biliary drainage and the common bile duct was intermittently sutured with 4-0 vicryl sutures.
  Arms: T-tube drainage

SUMMARY:
Residual and recurrent stones remain one of the most important challenges of hepatolithiasis which is reported in 20% to 50% of patients treated with these therapies. Up to now the most two common surgical procedures performed were choledochojejunostomy and T tube drainage as biliary drainage in hepatolithiasis. The goal of the present study was to evaluate the therapeutic safety, and perioperative and long-term outcomes of choledochojejunostomy versus T tube drainage for hepatolithiasis with sphincter of Oddi laxity.

DETAILED DESCRIPTION:
Background: SOL results in reflux of duodenal fluid and enteric bacteria infection, which lead to the formation of stones in the biliary tract. Roux-en-Y hepaticojejunostomy (HJ) shows considerable advantage for prevention of reflux of intestinal content into the bile duct. As a result, A randomized controlled trial (RCT) evaluate the therapeutic safety, and perioperative and long-term outcomes of HJ versus T tube drainage for hepatolithiasis with SOL.

Intervention: In total, 210 patients who met the following eligibly criteria were included and were randomized to choledochojejunostomy arm or T tube drainage in a 1:1 ratio.

Clinical data include: the incidence of biliary complications (stone recurrence; biliary stricture; cholangitis); sphincter of oddi function; biliary leakage; mortality; hepatic injury; quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age age between 18 and 70 years
2. Diagnosed as hepatolithiasis with sphincter of oddi laxity during operation
3. Achieved removing the focus, extraction of stones and correction of stricture during the operation
4. Written Informed consent
5. Willingness for complete 3-year follow-up.

Exclusion Criteria:

1. Participation in concurrent intervention trials with interference of outcome of this study
2. Associated tumor
3. Diagnosed as sphincter of oddi complete loss of function or normal
4. Underwent choledochojejunostomy at past
5. Lack of compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
stone recurrence rate | 3 years
  A recurrence stone was defined as a stone detected more than 3 months after surgery by any diagnostic method. (%)
biliary stricturer rate | 3 years
  Biliary stricture defined as clinically evident stenosis and subclinical stenosis proved by endoscopic examination or reoperation (%)
Cholangitis rate | 3 years
  The diagnosis of cholangitis is based on clinically evident (abdominal discomfort/pain, jaundice or fever associated with hepatolithiasis (%)

SECONDARY OUTCOMES:
sphincter of oddi function | an expected average of 120 minutes
  Grading criteria for the SO function were as follows: Normal; Laxity and Loss of function
Mortality | 90 days
  Operative mortality was defined as any death resulting from a complication during surgery
Biliary leakage | 90 days
  Biliary leakage was documented in line with the International Study Group of Liver Surgery (ISGLS) definitions and grading systems
total bilirubin | 90 days
  serum total bilirubin on 3 postoperative day (umol/L)
quality of life grading | 3 years
  Quality of life will be assessed by Visick score (Ⅰ～Ⅳ).

CONTACTS AND LOCATIONS:
Overall Officials: Bao Fu Liu, PhD, Study Chair — The First Affiliated Hospital of Anhui Medical University

REFERENCES:
- [Derived] Chen JM, Yan XY, Zhu T, Chen ZX, Zhao YJ, Xie K, Liu FB, Geng XP. T-tube drainage versus choledochojejunostomy in hepatolithiasis patients with sphincter of Oddi laxity: study protocol for a randomized controlled trial. Trials. 2020 Jun 29;21(1):586. doi: 10.1186/s13063-020-04483-z. PMID 32600474